CLINICAL TRIAL: NCT02902835
Title: BUPrenorphine Facilitated Access and Supportive Treatment--AIM 3
Brief Title: BUPrenorphine Facilitated Access and Supportive Treatment --AIM 3
Acronym: BUPFAST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant Funding Ended
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Aaron D. Fox, Assistant Professor of Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6559; K23DA034541 (NIH)
Record Dates: First submitted 2016-08-12; First posted 2016-09-16 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Opioid-related Disorders
Keywords: Buprenorphine treatment; Incarceration; Linkage Intervention; Opioid use disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Referral to treatment (Control) (Active Comparator): The control group will receive a referral to buprenorphine treatment by the research staff.
  Interventions: Behavioral: Referral to treatment
- BUP-FAST Intervention (Experimental): Thirty-six participants will each be paired with a trained peer mentor who will provide the BUP-FAST intervention.
  Interventions: Behavioral: BUP_FAST

INTERVENTIONS:
Behavioral: BUP_FAST — Peer mentorship including: buprenorphine education, identifying buprenorphine providers, accompaniment at appointments, and psychosocial support (via outreach phone calls)
  Arms: BUP-FAST Intervention
Behavioral: Referral to treatment — Participants will receive a pamphlet describing the buprenorphine treatment program at a Montefiore community health center.
  Arms: Referral to treatment (Control)

SUMMARY:
The goal of this study is to test whether peer mentors (i.e., individuals with past opioid addiction and prior incarceration) can facilitate entrance into buprenorphine (Suboxone) treatment for individuals with opioid use disorder who were recently released from jail or prison. In order to test whether it is helpful to have peer mentors paired with recently released individuals, the investigators will conduct an 18 month study, recruiting 72 formerly incarcerated individuals and assigning them by chance selection (like flipping a coin) to either a group that will receive peer mentorship or a group that will receive a referral to a community clinic.

DETAILED DESCRIPTION:
BUPrenorphine Facilitated Access and Supportive Treatment (BUP-FAST) is a peer mentorship intervention in which trained peer mentors will link formerly incarcerated individuals with opioid use disorder to addiction treatment (i.e. buprenorphine maintenance treatment) following release from incarceration. The current study is a pilot randomized control trial evaluating the effectiveness and feasibility of the peer mentorship intervention.

The investigators are conducting this study due to the high rates of relapse to opioid use following release from prison (up to 75% within 3 months) and difficulty that some formerly incarcerated individuals report in accessing effective treatments for opioid use disorder. The investigators hypothesize that having peer mentors - who themselves have experienced incarceration and have had success with buprenorphine treatment for opioid use disorder - assisting formerly incarcerated individuals in seeking treatment will result in higher rates of linkage to care in comparison to referral to a community health center for buprenorphine treatment.

In this 18-month randomized control trial of the BUP-FAST intervention, the investigators will recruit 72 formerly incarcerated individuals with opioid use disorder; half will then be randomized to receive the BUP-FAST intervention (peer mentorship); and the other half (control) will receive referral to a community health center for assessment for buprenorphine treatment. Medication will not be provided as part of this study. Participants will only receive buprenorphine treatment if they meet appropriate medical criteria after assessment at the community health center.

ELIGIBILITY:
Inclusion Criteria:

1. Current or prior (at the time of incarceration) opioid use disorder by DSM-V criteria
2. ≥ 18 years old
3. Fluent in English or Spanish
4. Released from incarceration in the last 4 weeks

Exclusion Criteria:

1. Current buprenorphine or methadone maintenance treatment
2. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Initiation of buprenorphine treatment | At 180 days post enrollment
  Initiation of buprenorphine treatment within 180 days of study enrollment will be confirmed by reviewing the patient's medical records. Participants will sign a release for protected health information in order to confirm buprenorphine induction and visits. Initiation of buprenorphine treatment will be defined as receiving one or more prescription for buprenorphine or buprenorphine-naloxone.

SECONDARY OUTCOMES:
Opioid use (self-reported) | At 45 days post enrollment
  Participants will complete interviews (adapted Addiction Severity Index) at study enrollment and at 45 days follow-up, self-reporting opioid use (heroin, opioid analgesics, methadone, illicit buprenorphine).
Opioid use (urine drug testing) | At 45 days post enrollment
  Participants will complete urine drug testing at study enrollment and at 45 days follow-up, assessing for any opioid use (opiates, oxycodone, methadone, buprenorphine).
Criminal activity | At 45 days post enrollment
  Participants will complete interviews (Addiction Severity Index) at study enrollment and 45 days follow-up, self-reporting involvement in criminal activities in the previous 30 days (# days with involvement).

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No